CLINICAL TRIAL: NCT05026255
Title: Assessment of Preload Dependency Via Measurement of Peripheral Venous Pressure During an Alveolar Recruitment Manoeuvre
Acronym: PVP-StepPEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment due to COVID 19
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A02683-36
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Intensive Care Patients

STUDY DESIGN:
Intervention Model Description: Prospective multicentre open-label study of mechanically ventilated intensive care patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mechanically ventilated intensive care patients. (Experimental): Observational data collected for patients in intensive care under mechanical ventilation.
  Interventions: Procedure: alveolar recruitment manoeuvre by pressure step

INTERVENTIONS:
Procedure: alveolar recruitment manoeuvre by pressure step — The application of alveolar recruitment manoeuvres consists of transiently increasing alveolar pressure in order to re-open collapsed alveolar territories and to re-ventilate poorly ventilated or non-ventilated lung areas.

SUMMARY:
Assessment of preload dependency via measurement of peripheral venous pressure during an alveolar recruitment manoeuvre.

Prospective multicentre open-label study of mechanically ventilated intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, for whom the trusted person designated by the patient or, failing that, a relative has read and signed the consent form for participation in the study
* Patient hospitalised in intensive care, under sedation and controlled mechanical ventilation
* Equipped with a central venous line in the superior vena cava territory and an arterial catheter.
* Whose state of health justifies vascular filling

Exclusion Criteria:

* Patient under legal protection, guardianship or curatorship
* Pregnant or breastfeeding woman
* Patient not affiliated to the French social security system
* Contraindication to the realization of an alveolar recruitment maneuver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure | through study completion, an average of 12 hours
  The correlation between the pairs of values of CVP and PVP during an alveolar recruitment manoeuvre will be evaluated by Pearson's coefficient or Spearman's coefficient if the distribution of the values is not parametric. The coefficient of determination r² will be calculated by linear regression between the 2 variables. Finally, the agreement between the two measurements will be evaluated by the Bland-Altman method: the Bland-Altman graph will be provided and the 95% agreement limits will be calculated (+/- 1.96 SD, SD being the standard deviation of the difference between the measurements).

SECONDARY OUTCOMES:
Secondary outcome measure | through study completion, an average of 12 hours
  Predictive value of the evolution of PVP during the recruitment manoeuvre: the ROC curve (receiver-operating characteristic) will be performed by logistic regression. The area under the ROC curve will be given as well as the sensitivity, specificity and negative and positive predictive values (Younden index will be used to determine the optimal threshold of PVP).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé de la Loire, Saint-Etienne, France